CLINICAL TRIAL: NCT04682327
Title: Observational Study on the Relationship Between Gut Microbiota and Immunotherapy Response of Non-small Cell Lung Cancer
Brief Title: Gut Microbiota and Cancer Immunotherapy Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2020-300
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responder group: After the 4 cycles of anti-PD-1/PD-L1 mAbs treatment, the investigators evaluated the subjects' response to anti-PD-1/PD-L1, according to the Response Evaluation Criteria In Solid Tumors (RECIST V1.1) or Modified RECIST 1.1 for immune based therapeutics (iRECIST) .
  Responders are defined as complete remission, partial remission, or stable disease.
  Interventions: Other: Response to anti-PD-1/PD-L1
- Nonresponder group: After the 4 cycles of anti-PD-1/PD-L1 treatment, the investigators evaluated the subjects' response to anti-PD-1/PD-L1, according to the Response Evaluation Criteria In Solid Tumors (RECIST V1.1) or Modified RECIST 1.1 for immune based therapeutics (iRECIST) .
  Nonresponders are defined as disease progression.
  Interventions: Other: Non-response to anti-PD-1/PD-L1

INTERVENTIONS:
Other: Response to anti-PD-1/PD-L1 — Response to anti-PD-1/PD-L1, after 4 cycles of anti-PD-1/PD-L1 treatment.
  Groups: Responder group
Other: Non-response to anti-PD-1/PD-L1 — Non response to anti-PD-1/PD-L1, after 4 cycles of anti-PD-1/PD-L1 treatment.
  Groups: Nonresponder group

SUMMARY:
This study will analyze the composition and diversity of the gut microbiota of patients with locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) through metagenomic high-throughput sequencing methods, and explore the relationship between the gut microbiota and anti-PD-1/PD-L1 treatment response.

This study will further understand the influence and mechanism of the gut microbiota on tumor immunotherapy, and will provide new ideas and theoretical basis for improving the efficacy of tumor immunotherapy by targeting the gut microbiota in the clinic, and benefit more NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this trial, fully understand this trial, and sign the Informed Consent Form (ICF).
2. 18-75 years old on the day of signing the ICF.
3. Locally advanced/metastatic non-small cell lung cancer diagnosed by histology or cytology. no epidermal growth factor receptor (EGFR) sensitive mutations, anaplastic lymphoma kinase (ALK) gene rearrangement, ROS Proto-oncogene 1 (ROS1) gene fusion.
4. receive anti-PD-1/PD-L1 for first-line treatment.
5. Have not received systemic treatment for locally advanced/metastatic NSCLC.
6. Have measurable target lesions judged by the investigator according to Response Evaluation Criteria In Solid Tumors (RECIST V1.1).
7. 0~1 ECOG score.
8. Life expectancy ≥ 12 weeks.
9. Have sufficient organ function, evaluated based on blood routine, renal function, liver function, and coagulation laboratory test results (and have not received blood transfusion or infusion of apheresis components within 14 days before the study drug administration , Erythropoietin, granulocyte colony stimulating factor and other medical support treatments).
10. Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within 7 days before the first medication, and the result is negative; WOBCP or men and their WOBCP partners should agree from signing the ICF to the last one. Take effective contraceptive measures within 6 months after taking the study drug.

Exclusion Criteria:

1. Before the first administration of the trial treatment: a) have received previous systemic cytotoxic chemotherapy for metastatic disease; b) have received other targeted or biological anti-tumor therapy for metastatic disease ; c) received major surgery (<3 weeks before the first dose); d) received lung radiotherapy >30 Gy within 6 months before the first dose of the trial treatment; e) the first trial treatment Palliative radiotherapy was completed within 7 days before administration.
2. Any other form of anti-tumor therapy is expected during the study period.
3. Live virus vaccines have been vaccinated within 30 days before the planned treatment. Seasonal influenza vaccine without live virus is allowed.
4. A history of past malignant disease is known, unless the subject receives potentially curative treatment and there is no evidence of disease recurrence within 5 years after starting treatment.
5. Accompanying known active central nervous system (CNS) metastasis and/or cancerous meningitis.
6. According to the standard of Common Adverse Event Terminology (CTCAE) 4th edition, peripheral neuropathy has been ≥2 grade.
7. Severe hypersensitivity reactions to other monoclonal antibody treatments have occurred in the past.
8. Accompanied by active autoimmune diseases, systemic treatment (ie, use of disease modifiers, corticosteroids or immunosuppressive drugs) is required within the past 2 years.
9. Are receiving long-term systemic steroid therapy. Subjects with asthma who require intermittent use of bronchodilators, inhaled steroids, or topical steroid injections are not excluded.
10. Have received any other anti-PD-1 or PD-L1 or PD-L2 drugs or antibodies in the past, or small molecule therapy that targets other immunomodulatory receptors or mechanisms. Participated in any other anti-PD-1/PD-L1 trials and received anti-PD-1/PD-L1 treatment. Such antibodies include (but are not limited to) antibodies against IDO, PD-L1, IL-2R and GITR.
11. Active infections requiring treatment.
12. Known human immunodeficiency virus (HIV) history (known HIV1/2 antibody positive). Accompanied by known active hepatitis B or C.
13. Being pregnant or breastfeeding, or expecting to conceive or conceive during the period of study drug treatment and within the required contraceptive period after the last administration of the study drug.
14. The researcher believes that there are any circumstances that are not suitable for selection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with local late/metastasis non-small cell lung cancer treated with the first-line treatment of anti-PD-1/PD-L1 treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Diversity and Composition of gut microbiota | At the end of Cycle 4 (each cycle is 21 days)
  The difference of gut microbiota diversity and composition between Responder group with Non-Responder group. Microbiota diversity will be quantified by α-diversity ( Faith's Phylogenetic Diversity) based on meta-genomics sequencing. Microbiota composition will be quantified by the operational taxonomic unit (OTU) in the stool.

SECONDARY OUTCOMES:
Concentration of peripheral blood mononuclear cells | At the end of Cycle 4 (each cycle is 21 days)
  The difference of composition and content of peripheral blood mononuclear cells (CD8+T-cells, NK cells and myelin-sourced inhibitory cells) between Responder group with Non-Responder group. The composition and content of CD8+T-cells, NK cells and myelin-sourced inhibitory cells were analyzed by flow cytometry.
Concentration of tumor immune related cytokines | At the end of Cycle 4 (each cycle is 21 days)
  The difference of the contents of tumor immune related cytokines (IFNγ、TNF、Granzyme A/B、Perforin and et al)between Responder group with Non-Responder group. The contents of tumor immune related cytokines were analyzed by enzyme-linked immunosorbent assay.
Incidence of anti-PD-1/PD-L1 related adverse events | through study completion, up to 2 years
  Number of patients with adverse events that received anti-PD-1/PD-L1 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xizhong Shen, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available from the principal investigator Taotao Liu at shen.xizhong@zs-hospital.sh.cn, beginning 6 months and ending 5 years after the trial results were published. The study protocol and statistical analysis plan are available online from https://clinicaltrials.gov/. All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 5 years after the trial results were published.
Access Criteria: All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
URL: http://clinicaltrials.gov/